CLINICAL TRIAL: NCT00868543
Title: Long or Very Long-Limb Gastric Bypass in Superobese
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaunas University of Medicine (Other)
Responsible Party: Almantas Maleckas, Kaunas University of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BE-2-37
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: Gastric bypass; obesity; superobese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long limb (Active Comparator): Hospitalized male or female subjects 18-65 years of age,obese with body mass index (BMI= kg/m²)>50.Patients without mental or nervous disorders interfering with adequate evaluation of one's health condition, who read the informed consent form and gave a written consent to participate in the study. Gastric bypass was performed with long (150 cm) alimentary Roux limb
  Interventions: Procedure: laparoscopic gastric Roux-en-Y gastric bypass
- Very long limb (Active Comparator): Hospitalized male or female subjects 18-65 years of age,obese with body mass index (BMI= kg/m²)>50.Patients without mental or nervous disorders interfering with adequate evaluation of one's health condition, who read the informed consent form and gave a written consent to participate in the study. Gastric bypass was performed with very long (250 cm) alimentary Roux limb
  Interventions: Procedure: laparoscopic gastric Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: laparoscopic gastric Roux-en-Y gastric bypass — The fundus is separated by linear cutter. The intestine is opened approximately 75 cm from the ligament of Treitz and approached to the stomach. The gastrojejunostomy is performed in antecolic position The jejunum has to be in an antimesenteric position. After removing the endocutter, the anastomotic incision is closed with a continuous suture. The distance between the gastrojejunostomy and jejunojejunostomy was measured on the antimesenteric border with the bowel on a stretch. The jejunojejunostomy is performed in 150cm distance from gastrojejunostomy. The anastomosis is made by a posterior staple line and an anterior suture line. Preparation of a small window for the endocutter branches into the jejunal mesenterium 2-3 cm proximal to the gastrojejunostomy and above the entero-intestinal anastomosis.
  Other Names: laparoscopic gastric bypass
  Arms: Long limb
Procedure: laparoscopic gastric Roux-en-Y gastric bypass — The fundus is separated by linear cutter. The intestine is opened approximately 75 cm from the ligament of Treitz and approached to the stomach. The gastrojejunostomy is performed in antecolic position The jejunum has to be in an antimesenteric position. After removing the endocutter, the anastomotic incision is closed with a continuous suture. The distance between the gastrojejunostomy and jejunojejunostomy was measured on the antimesenteric border with the bowel on a stretch. The jejunojejunostomy is performed in 250cm distance from gastrojejunostomy. The anastomosis is made by a posterior staple line and an anterior suture line. Preparation of a small window for the endocutter branches into the jejunal mesenterium 2-3 cm proximal to the gastrojejunostomy and above the entero-intestinal anastomosis.
  Other Names: laparoscopic gastric bypass
  Arms: Very long limb

SUMMARY:
The goal of this study is to compare the clinical efficacy (weight loss and metabolic changes) of long (150 cm) versus very long (250cm) Roux alimentary limb gastric bypass in superobese (BMI>50) patients.

DETAILED DESCRIPTION:
The study is a multicentre trial in which superobese (BMI>50) patients will be randomly assigned (in a 1:1 ratio) for laparoscopic gastric Roux-en-Y gastric bypass with: a) long (150 cm) or b) very long (250cm) alimentary Roux limb. Patients will be included from three hospitals: Kaunas University of Medicine Hospital (Lithuania), Klaipeda District Hospital (Lithuania), Vaasa Central Hospital (Finland) ) where preoperative investigation, the same technique surgical procedures and follow up will be performed acording approved protocol.

Approximate duration of subject participation

Subjects in the study will participate for approximately 5 years:

* Preoperative investigation and surgery 3- 5 days in the hospital;
* First follow up visit: 6 months after surgery;
* Next follow up visits: 12, 24, 36, 48 months after surgery;
* Last follow up visit: 5 years after surgery.
* The interim results after 12, 24 and 36 months will be calculated and presented before end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female subjects 18-65 years of age.
* Obese subjects with body mass index (BMI= kg/m²)>50
* Patients without mental or nervous disorders interfering with adequate evaluation of one's health condition.
* Patients who read the informed consent form and gave a written consent to participate in the study.

Exclusion Criteria:

* Previous open abdominal surgery, except appendectomy, cholecystectomy and gynaecological procedures.
* Presence of any significance cardiac, hepatic, renal, blood, alimentary tract disease which may lead to system or organ failure in intraoperative or postoperative period.
* Pregnant women.
* Subjects taking immunosuppressive therapy.
* Any concomitant condition that, in the opinion of the investigator, would preclude an operation and postoperative follow up acording to a protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
weight loss- we will compare percentage of excess body weight loss (%EWL) between groups. | 7 years

SECONDARY OUTCOMES:
To compare body mass index changes and absolute weight loss. To evaluate obesity-related medical problems. To obtain data about impromvement of metabolic syndrom. To compare quality of life changes between treatment arms. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Almantas Maleckas, Principal Investigator — Kaunas University of Medicine
Locations (1):
- KMUK, surgery department, Kaunas, Lithuania